CLINICAL TRIAL: NCT06273319
Title: The Effect of Oxygen Administration With Double Nasal Cannula on Respiratory Complications in Endoscopies
Brief Title: The Effect of Oxygen Application With Double Nasal Cannula on Respiratory Complications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, DUYGU DEMİROZ, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 010656
Record Dates: First submitted 2024-01-12; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Gastric Disease; Gastric Distress
Keywords: Desaturation; oxygen therapy; Sedoanalgesia
MeSH Terms: conditions — Stomach Diseases | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Patients who will receive 15 litres oxygen therapy (Placebo Comparator): : Patients who will receive 15 litres oxygen therapy, will be applied throughout the transaction.Patient saturation and complications such as bronchospasm and laryngospasm respiratory arrest will be recorded throughout the procedure.
  Interventions: Drug: OXYGEN THERAPY
- Group 2: Patients who will receive 30 litres oxygen therapy (Active Comparator): Patients who will receive 30 litres oxygen therapy,will be applied throughout the transaction.Patient saturation and complications such as bronchospasm and laryngospasm respiratory arrest will be recorded throughout the procedure.
  Interventions: Drug: OXYGEN THERAPY

INTERVENTIONS:
Drug: OXYGEN THERAPY — 15 AND 30 LT OXYGEN TREATMENT

SUMMARY:
To compare desaturation and respiratory complications by applying oxygen therapy with double nasal cannula to patients who are planned to undergo gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Two groups of patients scheduled for gastrointestinal endoscopy will be compared in terms of desaturation and respiratory complications by applying 15 litres of oxygen therapy to the first group and 30 litres to the second group with double nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

18-65 years old

PATIENTS WHO WILL HAVE ENDOSCOPY AND OR COLONOSCOPY

Exclusion Criteria:

* Chronic obstructive pulmonary disease Having low saturation Lung cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the amount of oxygen to prevent the peripheral oxygen saturation of the patients from falling below 95% | Up to 24 weeks
  Determination of the amount of oxygen to prevent the peripheral oxygen saturation of the patients from falling below 95%

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu universitesi, Malatya, Turkey (Türkiye)